CLINICAL TRIAL: NCT06609148
Title: Randomized, Double-Blind, Placebo-Controlled Trial of De Simone Formulation Probiotic in Patients With Bile Acid Malabsorption/Diarrhea Unassociated With Ileal Resection
Brief Title: Probiotic in Patients With Bile Acid Malabsorption/Diarrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Michael Camilleri, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24-003006
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Bile Acid Malabsorption; Bile Acid Diarrhea

STUDY DESIGN:
Intervention Model Description: Randomized controlled study of probiotic combination versus placebo in patients with bile acid diarrhea
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental)
  Interventions: Dietary Supplement: De Simone formulation probiotic
- Control Group (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: De Simone formulation probiotic — Subjects will be given De Simone formulation probiotic 900 billion CFU, 3 times per day for 21-24 days
  Arms: Probiotic Group
Dietary Supplement: Placebo — Subjects will be given a placebo for 21-24 days
  Arms: Control Group

SUMMARY:
The purpose of this study is to assess effect of the DSF probiotic on fecal bile acid levels in patients with BAM.

DETAILED DESCRIPTION:
In this placebo-controlled trial, the De Simone combination probiotic formulation will be tested in 12 patients in each treatment arm. The patient's will be previously diagnosed with bile acid diarrhea. The objective is to assess the effects of this probiotic on fecal blood low acid levels in patients with bile acid diarrhea. Secondary objectives are to evaluate changes in% primary fecal bile acids in a single stool sample, serum 7 alpha C4, intestinal permeability, stool consistency and frequency, fecal short chain fatty acids, and fecal micro biome composition and diversity

ELIGIBILITY:
Inclusion criteria:

* Prior diagnosis of bile acid malabsorption documented in the medical history based on

  * either serum C4 >52.5ng/mL, or
  * fecal 48h total BA excretion >2337 μmol/48h, or
  * primary BA >5% 48h stool collection or >10% in single stool sample.
* 7-day stool dairy with an average stool consistency based on the Bristol Stool Form Scale, BSFS, with a grade greater than 5. Note: If Inclusion criteria 3 is not met, participants may choose to have their blood drawn clinically to further determine eligibility.
* For women of childbearing potential

  * A negative urine pregnancy test prior to dispensing the study product
  * Agreement to comply with approved methods of contraception during the whole study: unless they meet the criteria of post-menopausal, i.e. 12 months of spontaneous amenorrhea, women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner, should use one or more of the following acceptable methods of contraception that should be maintained throughout the study:

    * Surgical sterilization
    * Hormonal contraception (implantable, patch, oral, intra-muscular)
    * Intra-uterine device
    * Double barrier method (diaphragm plus condom)
    * At the discretion of the investigator, total abstinence is acceptable in cases where age, career, lifestyle, or sexual orientation of the patient ensures compliance

Exclusion criteria:

* Use of oral antibiotics and probiotics within the last 4 weeks.
* Pregnancy or lactation.
* Concomitant use of bile acid sequestrants, must stop 10 days before starting 7-day stool dairy and for the duration of the study.
* History of ileal resection.
* Diabetes mellitus (type 1)
* BMI ≥ 40 kg/m^2
* Diagnosis of gastrointestinal diseases that are associated with inflammation such as inflammatory bowel diseases and celiac diseases or gastrointestinal infection in the prior 4 weeks
* Any condition or personal circumstance that, in the opinion of the investigator, renders the subject unlikely or unable to comply with the full study protocol or could interfere with the study assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-01-02 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Change in fecal bile acid concentration | Baseline, 24 days
  Reported as micromoles per g stool and % primary bile acids

SECONDARY OUTCOMES:
Change in intestinal permeability | Baseline, 24 days
  Intestinal permeability will be measured using the standardized, validated 13C-mannitol and lactulose urine excretion test and reported as a ratio of the percentage excretion of lactulose and mannitol in urine

OTHER OUTCOMES:
Changes in symptoms based on daily stool diary acquired for 7 days' baseline and the 21 days of intervention | Baseline, 24 days
  The stool diary will measure stool consistency based on the Bristol Stool Form Scale (BSFS) from 1 to 7 where 7 is watery stool and 1 is hard stool and therefore a small number indicated a favorable outcome

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, DSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No